CLINICAL TRIAL: NCT02443376
Title: The Effects of Hemodialysis Session on Pulse Wave Velocity and Central Arterial Pressure
Brief Title: The Effects of Hemodialysis Session on Vascular Stiffness
Acronym: PWV/CP/HD
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Czyżewski, Lukasz Czyzewski, Medical University of Warsaw
Other Study IDs: PWV/CP/HD/2015/05
Record Dates: First submitted 2015-05-10; First posted 2015-05-13 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Arteriopathic Disease; Arterial Calcification; Complication of Hemodialysis; Aortic Stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hemodialysis patients: Stable end-stage renal disease patients on maintenance conventional hemodialysis received 4-5 hours of treatment thrice weekly. Pulse wave velocity and central aortic pressure was measured before and after the midweek dialysis session.Overhydration Urea distribution volume (V) Total body water, extracellular and intracellular water Lean Tissue Index (LTI) Fat Tissue Index (FTI) Body Cell Mass (BCM) was measured before the midweek dialysis session just after Complior device
  Interventions: Device: Complior Analyse System; Device: BCM- Body Composition Monitor
- Healthy subjects: Medical staff: medical doctors, nurses
  Interventions: Device: Complior Analyse System

INTERVENTIONS:
Device: Complior Analyse System — Pulse Wave Velocity PWV and central Pressure analysis
Device: BCM- Body Composition Monitor — BCM - Body Composition Monitor gives information about:
  Overhydration Urea distribution volume (V) Total body water, extracellular and intracellular water Lean Tissue Index (LTI) Fat Tissue Index (FTI) Body Cell Mass (BCM)
  Groups: Hemodialysis patients

SUMMARY:
Central blood pressure and pulse wave velocity were measured using a Complior Analyse device before and immediately after the end of the dialysis session.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* patients on maintenance hemodialysis at least 3 months
* stable dry weight
* single-pool Kt/V >1.4
* no clinical cardiovascular disease during the 6 months preceding entry
* medical staff (medical doctors, nurses)

Exclusion Criteria:

* not meet the above criteria
* episode of illness (for example: infection)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 80 consecutive patients on maintenance hemodialysis and 30 healthy subjects were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Differences in carotid-femoral pulse wave velocity [m/s] just before and after hemodialysis session | 1 day

SECONDARY OUTCOMES:
Differences in central aortic pressure [mmHg] just before and after hemodialysis session | 1 day
Differences in central aortic pressure [mmHg] and cuff blood pressure [mmHg] just before and after hemodialysis session | 1 day
Impact of fluid and nutritional status on carotid-femoral pulse wave velocity and central aortic pressure | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Wyzgał, Professor, Study Chair — Medical University of Warsaw, Department of Nephrologic Nursing
Locations (1):
- Medical University of Warsaw, Warsaw, Mazovian, Poland

REFERENCES:
- [Background] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Assessment of health-related quality of life of patients after kidney transplantation in comparison with hemodialysis and peritoneal dialysis. Ann Transplant. 2014 Nov 9;19:576-85. doi: 10.12659/AOT.891265. PMID 25382249
- [Result] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Comparative analysis of hypertension and its causes among renal replacement therapy patients. Ann Transplant. 2014 Nov 3;19:556-68. doi: 10.12659/AOT.891248. PMID 25365639
- [Result] Czyzewski L, Wyzgal J, Kolek A. Evaluation of selected risk factors of cardiovascular diseases among patients after kidney transplantation, with particular focus on the role of 24-hour automatic blood pressure measurement in the diagnosis of hypertension: an introductory report. Ann Transplant. 2014 Apr 28;19:188-98. doi: 10.12659/AOT.890189. PMID 24770703